CLINICAL TRIAL: NCT01277887
Title: Smoking Cessation for Smokers With Sleep Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1005006857; P50DA009241-16 (NIH)
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Nicotine Dependence; Cigarette Smoking; Insomnia
Keywords: Smoking; Nicotine; Nicotine polacrilex; Nicotine replacement
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Sleep Initiation and Maintenance Disorders; Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-Behavioral Counseling (Active Comparator): The intervention consists of 8 sessions provided over 10 weeks. Counseling commences 4 weeks before quitting smoking. Participants will also receive the nicotine patch for 6 weeks starting on the day of quit date.
  Interventions: Behavioral: Cognitive-Behavioral Counseling
- Smoking Cessation Counseling (Placebo Comparator): The intervention consists of 8 sessions provided over 10 weeks. Counseling commences 4 weeks before quitting smoking. Participants will also receive the nicotine patch for 6 weeks starting on the day of quit date.
  Interventions: Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Counseling — The cognitive-behavioral intervention integrates standard smoking counseling adapted from the American Lung Association Freedom from Smoking program along with cognitive-behavioral techniques for improving insomnia.
  Other Names: CBT-I + SC
  Arms: Cognitive-Behavioral Counseling
Behavioral: Smoking Cessation Counseling — The smoking cessation counseling intervention will incorporate standard psychoeducational and behavioral smoking counseling techniques adapted from the American Lung Association Freedom from Smoking program.
  Other Names: SC
  Arms: Smoking Cessation Counseling

SUMMARY:
This is a pilot research study examining two types of behavioral counseling along with the nicotine patch for smoking cessation. The study is designed to find out whether one of these counseling interventions is more effective for smoking cessation among individuals with sleep problems. The study has three parts: 1) an intake session; 2) a 10-week treatment phase, and 3) a 1-month follow-up.

DETAILED DESCRIPTION:
This is a developmental study to: 1) create and test an integrated cognitive-behavioral smoking cessation and insomnia intervention with 30 smokers who report current insomnia. Participants are randomized to 1 of 2 counseling conditions. The cognitive-behavioral intervention provides standard care smoking counseling along with counseling to address insomnia. The smoking counseling intervention provides standard care smoking counseling adapted from the American Lung Association Freedom from Smoking program. Efficacy data from this trial will be used to determine effect size estimates for biologically confirmed self-reported point prevalence smoking abstinence at the end of treatment and 1 month after completing treatment. Changes in sleep efficiency and self-control to resist smoking urges will also be examined. If the effect size estimates are sufficiently large and medically important to pursue a definitive trial, these data will be used to propose a full scale large study.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 75.
* Smoking 10 or more cigarettes per day for at least 1 year.
* An expired air breath carbon monoxide level > 10 ppm.
* Motivated to stop smoking.
* Understand English.
* Meet DSM-IV criteria for insomnia.
* Report sleep latency or waking after sleep onset >30 minutes on ≥6 occasions within past month.

Exclusion Criteria:

* History of allergic reactions to adhesives.
* Unstable psychiatric/medical conditions such as current suicidal or homicidal ideation, acute psychosis, dementia.
* Have a current diagnosis of DSM-IV alcohol or drug dependence other than nicotine.
* Use of tobacco products other than cigarettes or use of marijuana.
* Intention to use nicotine replacement therapy, varenicline, or bupropion during study participation.
* Females of childbearing potential who are pregnant, nursing, or not practicing effective contraception (oral, injectable, or implantable contraceptives, intrauterine device, or barrier method with spermicide).
* New onset of psychiatric disorders or new psychotropic medications within the past 3 months.
* Inability to read/understand English.
* History of sleep apnea based on responses to Berlin Questionnaire.
* History of restless leg syndrome.
* Current night or rotating shift work.
* Proposed travel across 2 or more time zones during study participation.
* Medical/psychiatric conditions contraindicated for sleep restriction (i.e., seizure disorders, severe excessive daytime sleepiness - Epworth Scale >18, and bipolar disorder).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fucito, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized between 9/2/11-12/6/11 at an outpatient research clinic.
Pre-assignment Details: Prior to randomization, inclusion and exclusion criteria were assessed. Reasons for exclusion included CBT-I contraindicated medical/psychiatric conditions, not meeting smoking criteria, other drug dependence, and not meeting sleep criteria.
Period: Pre-Quit Treatment Phase
Arm/Group | Cognitive-Behavioral Counseling | Smoking Cessation Counseling
Started | 9 | 10
Entered Study | 7 | 10
Completed | 6 | 10
Not Completed | 3 | 0
Not completed — No longer interested in treatment | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Post-Quit Treatment Phase
Arm/Group | Cognitive-Behavioral Counseling | Smoking Cessation Counseling
Started | 6 | 10
Completed | 3 | 5
Not Completed | 3 | 5
Not completed — No longer interested in treatment | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Counseling | Smoking Cessation Counseling | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.86 (15.07) | 51.20 (10.73) | 51.47 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: Smoking abstinence is operationally defined as "no smoking on the last 7 days of the last week of treatment. And no smoking within the last 7 days at the first follow-up visit 4 weeks after completing treatment."
Time Frame: 1 Week
Measure: Number; unit: participants
Arm/Group | Cognitive-Behavioral Counseling | Smoking Cessation Counseling
Number analyzed (Participants) | 7 | 10
participants
  7-day PPA at end of treatment | 1 | 2
  7-day PPA at follow up | 1 | 0

2. Secondary Outcome: Self-Control to Resist Smoking Cues
Description: To develop an effect size estimate for changes in self-control to resist smoking cues from baseline to the day before quitting smoking comparing smokers in the two counseling conditions.
Time Frame: 4 Weeks
Population: These data were not collected.
Arm/Group | Cognitive-Behavioral Counseling | Smoking Cessation Counseling
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Sleep Efficiency
Description: Self-reported sleep efficiency subscale of the Pittsburgh Sleep Quality Index. This is calculated as the percentage of total time spent asleep in a night compared to the total time spent in bed, multiplied by 100.
Time Frame: Change from Baseline at 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of time asleep in bed
Arm/Group | Cognitive-Behavioral Counseling | Smoking Cessation Counseling
Number analyzed (Participants) | 7 | 10
percentage of time asleep in bed
  Baseline | 85.10 (13.08) | 72.51 (15.43)
  Week 4 | 92.17 (11.90) | 77.56 (18.11)

ADVERSE EVENTS:
Arm/Group | Cognitive-Behavioral Counseling | Smoking Cessation Counseling
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 6/7 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive-Behavioral Counseling (N=7) | Smoking Cessation Counseling (N=10)
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Decreased Appetite (General disorders) | 1 | 3
Increased Appetite (General disorders) | 2 | 5
Headache (General disorders) | 2 | 1
Dizziness (General disorders) | 0 | 2
Rapid Heartbeat (Vascular disorders) | 0 | 3
Fatigue (General disorders) | 2 | 0
Nervousness/Anxiety (Psychiatric disorders) | 1 | 2
Insomnia (General disorders) | 2 | 0
Extreme Sleepiness (General disorders) | 2 | 2
Depression (Psychiatric disorders) | 1 | 3
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Vivid Dreams (General disorders) | 2 | 4
Sweating (Skin and subcutaneous tissue disorders) | 1 | 2
Bowel Changes- Increased Frequency (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Other (General disorders) | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes